CLINICAL TRIAL: NCT01470469
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Assess the Safety and Tolerability of SPD503 in Subjects Aged 6-17 Years With Generalized Anxiety Disorder (GAD), Separation Anxiety Disorder (SAD), or Social Phobia (SoP).
Brief Title: SPD503 in Subjects Aged 6-17 Years With Generalized Anxiety Disorder (GAD), Separation Anxiety Disorder (SAD), or Social Phobia (SoP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD503-210
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Generalized Anxiety Disorder (GAD); Anxiety, Separation; Phobia, Social
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety, Separation; Phobia, Social | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- SPD503 (Active Comparator)
  Interventions: Drug: SPD503 (extended-release Guanfacine hydrochloride)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD503 (extended-release Guanfacine hydrochloride) — Once-daily oral dosing of SPD503 in the evening ranging from 1-6 mg for 12 weeks (6 week dose optimization and 6 week dose maintenance).
  Other Names: Intuniv
  Arms: SPD503
Drug: Placebo — Once-daily oral dosing in the evening for 12 weeks.
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and tolerability of SPD503 in subjects aged 6-17 years with GAD, SAD, or SoP based on treatment emergent adverse events (TEAEs), vital signs and ECGs.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient subjects aged 6-17 years inclusive at the time of consent/assent (Screening Visit [Visit 1] only).
2. Subject's parent or legally authorized representative (LAR) must provide signature of informed consent, and there must be documentation of assent by the subject indicating that the subject is aware of the investigational nature of the study and the required procedures in accordance with the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guidance E6 (1996) and applicable regulations before completing any study-related procedures (Screening Visit [Visit 1] only).
3. Subject meets Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) criteria for a Primary Diagnosis of 1 or any combination of the following; GAD, SAD or SoP (300.02, 309.21 and 300.23), based on a detailed psychiatric evaluation at screening including completion of the Anxiety Disorders Interview Schedule for DSM-IV Child Version (ADIS-C).
4. Subject has a score of >/= 4 on the Clinician Severity Rating Scale for the Principal Diagnosis on the ADIS-C CSR) at the Screening Visit (Visit 1) and the Baseline Visit (Visit 2).
5. Subject is functioning at an age-appropriate level intellectually, as determined by the Investigator.
6. Subject and parent/LAR understand, are able, willing, and likely to fully comply with the study procedures and restrictions defined in this protocol, in the opinion of the Investigator.
7. Subject is able to swallow intact tablets.
8. Subjects who are females of child-bearing potential (FOCP), defined as >/= 9 years of age or if <9 years of age are post-menarchal, must have a negative serum beta Human Chorionic Gonadotropin (HCG) pregnancy test at the Screening Visit (Visit 1) and a negative urine pregnancy test at the Baseline Visit (Visit 2) and Week 12 (Visit 11/ET). Females of child-bearing potential must abstain from sexual activity that could result in pregnancy or agree to use acceptable methods of contraception.

Exclusion Criteria:

1. Subject has a current co-morbid psychiatric diagnosis of a major depressive disorder, bipolar illness, psychosis, a pervasive development disorder other than Asperger's Syndrome, attention deficit hyperactivity disorder, an eating disorder, or substance abuse disorder.
2. Subject has an ADIS-C CSR score for any Axis I disorder that is greater than the ADIS-C CSR score for their Principal Diagnosis of GAD, SAD, or SoP.
3. Subject has any condition or illness which, in the opinion of the Investigator, represents an inappropriate risk to the subject and/or could confound the interpretation of the study.
4. Within 14 days prior to the Baseline Visit subject has received any evidence-based psychosocial intervention intended to reduce anxiety symptoms i.e. Individual Cognitive Behavioral Therapy, Group Cognitive Behavioral Therapy, or Social Effectiveness Training.
5. Subject has started or changed the type or intensity of a non evidence-based psychosocial intervention intended to reduce anxiety symptoms within 6 weeks prior to the Baseline Visit (Visit 2).
6. Subject has a known history or presence of structural cardiac abnormalities, serious heart rhythm abnormalities, syncope, cardiac conduction problems (e.g., clinically significant heart block), exercise-related cardiac events including syncope and pre syncope, or clinically significant bradycardia.
7. Subject with orthostatic hypotension or a known history of controlled or uncontrolled hypertension.
8. Subject has a blood pressure measurement above the 95th percentile for age, sex, and height.
9. Subject has a history of a seizure disorder other than a single childhood febrile seizure occurring before the age of 3 years.
10. Subject is currently considered at risk for suicide in the opinion of the Investigator, has previously made a suicide attempt, or is currently demonstrating active suicidal ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the Investigator.
11. Subject is unable to limit caffeine intake to 2 servings per day throughout participation in the study beginning at time of informed consent/assent.
12. Subject has a history of alcohol or other substance abuse or dependence, as defined by DSM-IV within the last 6 months.
13. Clinically important abnormality on drug and alcohol screen at the Screening Visit (Visit 1) or Baseline Visit (Visit 2).
14. History of failure to respond to 2 adequate trials (consisting of an appropriate dose and adequate duration of therapy) of an SSRI or one trial of cognitive behavioral therapy for the treatment of GAD, SAD, or SoP.
15. Subject is well controlled on anxiolytic pharmacologic or non-pharmacologic therapy with acceptable tolerability.
16. Subject is currently using a prohibited medication or other medications, including herbal supplements that have identified anxiolytic or anxiogenic effects, that affect BP or heart rate or that have CNS effects in violation of the protocol-specified washout criteria at the Baseline Visit (Visit 2).
17. Subject is currently using valproic acid or any drug known to inhibit or induce CYP3A4/5 in violation of the protocol-specified washout criteria at the Baseline Visit (Visit 2).
18. Use of another investigational medicinal product or participation in a clinical study within 30 days prior to the Baseline Visit (Visit 2).
19. Subject is significantly overweight based on Center for Disease Control and Prevention body mass index (BMI)-for-age sex specific charts at the Screening Visit (Visit 1). Significantly overweight is defined as a BMI >95th percentile for this study.
20. Subject has a known or suspected allergy, hypersensitivity, or clinically significant intolerance to guanfacine hydrochloride or any components found in SPD503.
21. Subject is female and is pregnant or currently lactating.
22. Subject failed screening or was previously enrolled in this study.
23. Subject has another member of the same household currently participating in this study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2012-01-04 (Actual); Primary Completion 2013-07-15 (Actual); Study Completion 2013-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (33):
- United States (33):
  - Birmingham Research Group, Inc, Birmingham, Alabama
  - Dr. Joseph H. Rodd, Carson, California
  - Sun Valley Research, Imperial, California
  - Irvine Center for Clinical Research, Irvine, California
  - Sharp Mesa Vista Hospital, Clinical Research Department, San Diego, California
  - Elite Clinical Trials, Inc, Wildomar, California
  - Florida Clinical Research Center, Bradenton, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Kolin Research Group, Winter Park, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Institute of Behavioral Medicine, LLC, Smyrna, Georgia
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Midwest Research Group, Saint Charles, Missouri
  - Premier Psychiatric Group, LLC, Lincoln, Nebraska
  - Center for Psychiatry and Behavioral Medicine, Inc, Las Vegas, Nevada
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Columbia University, NY State Psychiatric Institute, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Duke University Medical Center, Duke Child and Family Study Center, Durham, North Carolina
  - University of Cincinnati, Department of Psychiatry and Behavioral Neuroscience, Cincinnati, Ohio
  - University Hospitals of Cleveland Medical Center, Cleveland, Ohio
  - Professional Psychiatric Services, Mason, Ohio
  - North Star Research, Middleburg Heights, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - FutureSearch Clinical Trials, LP, Austin, Texas
  - Houston Clinical Trials LLC, Houston, Texas
  - Ericksen Research and Development, Clinton, Utah
  - NeuroScience, Inc., Herndon, Virginia

REFERENCES:
- [Derived] Strawn JR, Compton SN, Robertson B, Albano AM, Hamdani M, Rynn MA. Extended Release Guanfacine in Pediatric Anxiety Disorders: A Pilot, Randomized, Placebo-Controlled Trial. J Child Adolesc Psychopharmacol. 2017 Feb;27(1):29-37. doi: 10.1089/cap.2016.0132. Epub 2017 Feb 6. PMID 28165762

RESULTS

PARTICIPANT FLOW:
Groups:
- SPD503: Once-daily oral dosing of SPD503 in the evening ranging from 1-6 mg for 12 weeks.
Period: Overall Study
Arm/Group | PLACEBO | SPD503
Started | 21 | 62
Completed | 11 | 38
Not Completed | 10 | 24
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Lack of Efficacy | 1 | 7
Not completed — Adverse Event | 0 | 7
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Other | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PLACEBO | SPD503 | Total
Number analyzed (Participants) | 21 | 62 | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.8 (3.46) | 11.7 (3.39) | 11.7 (3.38)
Age, Customized [Count of Participants; unit: Participants]
  Age 6-12 years | 12 | 38 | 50
  Age 13-17 years | 9 | 24 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 38 | 48
  Male | 11 | 24 | 35
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 21 | 62 | 83

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Systolic Blood Pressure at Up to 12 Weeks
Time Frame: Baseline and up to 12 weeks
Population: Safety Analysis Set consisted of all subjects who had taken at least 1 dose of investigational product and had at least 1 post-dose safety assessment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 19 | 59
mmHg | -1.7 (11.18) | -2.3 (11.40)

2. Primary Outcome: Change From Baseline in Diastolic Blood Pressure at Up to 12 Weeks
Time Frame: Baseline and up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 19 | 59
mmHg | 0.9 (7.37) | -1.3 (9.09)

3. Primary Outcome: Change From Baseline in Pulse Rate at Up to 12 Weeks
Time Frame: Baseline and up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 19 | 59
beats/min | -0.5 (11.09) | -1.8 (11.54)

4. Primary Outcome: Change From Baseline in Height at up to 12 Weeks
Time Frame: Baseline and up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 19 | 59
cm | 0.5 (0.91) | 1.0 (1.79)

5. Primary Outcome: Change From Baseline in Weight at up to 12 Weeks
Time Frame: Baseline and up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 19 | 59
kg | 0.7 (1.73) | 1.3 (1.57)

6. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) QRS Interval at up to 12 Weeks
Description: QRS complex is a portion of the ECG tracing that represents depolarization of the ventricular myocardium.
Time Frame: Baseline and up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 19 | 55
msec | 0.7 (6.50) | 0.1 (5.33)

7. Primary Outcome: Change From Baseline in ECG QTcF Interval at up to 12 Weeks
Description: The QT interval is the time from the start of the Q wave to the end of the T wave. It is a portion of the ECG tracing that represents the time taken for ventricular depolarisation and repolarisation. The QTcF includes a correction factor to help account for changes in heart rate.
Time Frame: Baseline and up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | PLACEBO | SPD503
Number analyzed (Participants) | 19 | 55
msec | 0.3 (9.38) | 4.1 (14.01)

ADVERSE EVENTS:
Arm/Group | PLACEBO | SPD503
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/62
Other Adverse Events (participants affected / at risk) | 10/21 | 48/62
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=21) | SPD503 (N=62)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 10 (17)
Constipation (Gastrointestinal disorders) | 0 (0) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 5 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 6 (7)
Fatigue (General disorders) | 0 (0) | 13 (16)
Irritability (General disorders) | 1 (1) | 4 (4)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (3)
Joint sprain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 6 (6)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 7 (8)
Dizziness postural (Nervous system disorders) | 0 (0) | 7 (11)
Headache (Nervous system disorders) | 4 (7) | 22 (26)
Sedation (Nervous system disorders) | 2 (2) | 6 (7)
Somnolence (Nervous system disorders) | 1 (2) | 17 (30)
Initial insomnia (Psychiatric disorders) | 1 (1) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
Efficacy endpoints were exploratory. No statistical testing was performed because the study was not powered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.